CLINICAL TRIAL: NCT04644497
Title: Comparison of Different Anterior Cruciate Ligament Surgery Techniques in Skeletally Immature Patients.
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Other Study IDs: EC 1-10-72-246-20
Record Dates: First submitted 2020-11-16; First posted 2020-11-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transphyseal drilling technique
  Interventions: Procedure: ACL-reconstruction
- Physeal sparing drilling technique
  Interventions: Procedure: ACL-reconstruction

INTERVENTIONS:
Procedure: ACL-reconstruction — Surgery technique in skeletally immature patients

SUMMARY:
This cohort study compares to groups of patients with reconstruction of anterior cruciate ligament (ACL). Patients in group 1 had ACL-reconstruction in the years 2001-2010 with a transphyseal drilling technique. Patient in group 2 had ACL-reconstruction in the years 2013-2018 with a physeal sparing technique.

Data including: x-ray exam, patient reported questionnaires and clinical evaluation will be compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* ACL reconstruction as skeletally immature

Exclusion Criteria:

* Other ligament injuries in index knee
* Other ligament injuries in opposite knee
* Revision ACL reconstruction
* Pregnant
* Not able to read or understand the danish languages

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population:
  -ACL-reconstruction in one knee, operated in to periods (2001-2010 or 2013-2018) with two different techniques in each period.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Leg-length differences | 2 Years Follow-up
  X-ray evaluation
Knee Angle differences | 2 Years Follow-up
  X-ray evaluation

SECONDARY OUTCOMES:
Knee Laxity | 2 Years Follow-up
  Clinical evaluation with rolimeter (arthrometer)
IKDC-Questionnaire | 2 Years Follow-up
  The International Knee Documentation Committee (IKDC Questionnaire)
Tegner-Questionnaire | 2 Years Follow-up
  Tegner (Activity function score)
KOOS- Questionnaire | 2 Years Follow-up
  Knee injury and Osteoarthritis Outcome Score (KOOS)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No